CLINICAL TRIAL: NCT01585324
Title: Open, Multicenter Phase IV Study, Evaluating Drop of Hemoglobin in Association to the Rate of Sustained Virological Response in Chronic Hepatitis C Patients Treated With Ribavirin (Copegus®) in Combination With Standard Treatment (ANECO)
Brief Title: A Study of The Relationship Between Drop in Hemoglobin and Sustained Virological Response in Patients With Chronic Hepatitis C Treated With Copegus (Ribavirin) and Pegasys (Peginterferon Alfa-2a)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25186; 2011-001256-10 (EudraCT Number)
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg subcutaneously weekly
Drug: ribavirin [Copegus] — 1000 mg or 1200 mg orally daily

SUMMARY:
This open-label, multicenter, phase IV study will evaluate the relationship between the drop in hemoglobin levels and sustained virological response in patients with chronic hepatitis C genotype 1 treated with Copegus (ribavirin) and Pegasys (peginterferon alfa-2a). Patients will receive Copegus 1000 mg or 1200 mg orally daily and Pegasys 180 mcg subcutaneously weekly. Anticipated time on study treatment, depending on virological response, will be 48 or 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis C, genotype 1
* Treatment-naïve or patients who relapsed or failed to respond to previous combination therapy with interferon and ribavirin
* Detectable HCV-RNA
* Fertile males and females of child-bearing potential must agree to use two forms of contraception during treatment and for 6 months after treatment end

Exclusion Criteria:

* Pregnant or breast-feeding women
* Male partners of pregnant women
* History or evidence of a medical condition associated with chronic liver disease other than HCV
* Co-infection with active hepatitis A, hepatitis B and/or HIV virus
* Hepatocellular carcinoma
* History or evidence of oesophageal varices or other conditions consistent with decompensated liver disease
* Anemia
* Any patient with increased baseline risk for anemia (e.g. thalassemia, spherocyctosis, history of GI bleeding)
* History or evidence of significant cardiovascular disease
* Kidney disease
* Severe retinopathy
* History of severe psychiatric disease, especially depression
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) </= 6 months prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Most, Czechia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This clinical trial was originally planned to be conducted in 4 clinical trial centers in the Czech Republic. However, due to failure in manufacturing of the drug Pegasys, 3 of the previously approved study centers withdrew from participation. Consequently, the sponsor decided to conduct the clinical trial in 1 of the 4 originally planned centers.
Groups:
- Peginterferon Alpha-2a + Ribavirin: Participants infected with hepatitis C virus (HCV) genotype 1, who were either treatment naïve or failed to respond to previous combination therapy with interferon and ribavirin, were included in the study. These participants were treated with a combination therapy of peginterferon alpha-2a injection at a dose of 180 micrograms (mcg) subcutaneously once a week and ribavirin tablet, 1000-1200 milligrams (mg) by body weight (1000 mg if weight less than (<) 75 kilogram [kg]; 1200 mg if weight greater than or equal to (≥) 75 kg) orally split into 2 daily doses, for a total of 48 weeks.
Period: Overall Study
Arm/Group | Peginterferon Alpha-2a + Ribavirin
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Peginterferon Alpha-2a + Ribavirin: Participants infected with HCV genotype 1, who were either treatment naïve or failed to respond to previous combination therapy with interferon and ribavirin, were included in the study. These participants were treated with a combination therapy of peginterferon alpha-2a injection at a dose of 180 mcg subcutaneously once a week and ribavirin tablet, 1000-1200 mg by body weight (1000 mg if weight <75 kg; 1200 mg if weight ≥75 kg) orally split into 2 daily doses, for a total of 48 weeks.
Arm/Group | Peginterferon Alpha-2a + Ribavirin
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response (SVR) 24 Weeks After End of Treatment
Description: SVR was defined as a disappearance of HCV viral load 24 weeks after the end of the treatment.
Time Frame: 24 weeks after the end of treatment (72 weeks)
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alpha-2a + Ribavirin
Number analyzed (Participants) | 30
percentage of participants | 83.3 [65.28 to 94.36]
Statistical Analysis 1: Comparison: Peginterferon Alpha-2a + Ribavirin; Test type: Superiority or Other; p = 0.8333, ANCOVA; The analysis of covariance (ANCOVA) test for the efficacy of SVR achievement (Yes/No), treatment adjustment and baseline hemoglobin value was used

2. Primary Outcome: Change From Baseline in Hemoglobin Level at Week 12 of Treatment Among Participants With or Without SVR
Description: Change in hemoglobin level from a baseline level was assessed in the group of participants who achieved SVR and in the group of participants without SVR.
Time Frame: Baseline and Week 12
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Groups:
- Participants With SVR: Included all participants infected with HCV genotype 1, who were either treatment naïve or failed to respond to previous combination therapy with interferon and ribavirin, but achieved SVR after treatment with a combination therapy of peginterferon alpha-2a at a dose of 180 mcg subcutaneously once a week and ribavirin 1000-1200 mg by body weight (1000 mg if weight <75 kg; 1200 mg if weight ≥75 kg) orally once daily in 2 divided doses, for a total of 48 weeks. SVR response was defined as a disappearance of HCV viral load 24 weeks after the end of the treatment.
- Participants Without SVR: Included all participants infected with HCV genotype 1, who were either treatment naïve or failed to respond to previous combination therapy with interferon and ribavirin, and did not achieve SVR after treatment with a combination therapy of peginterferon alpha-2a at a dose of 180 mcg subcutaneously once a week and ribavirin 1000-1200 mg by body weight (1000 mg if weight <75 kg; 1200 mg if weight ≥75 kg) orally once daily in 2 divided doses, for a total of 48 weeks. SVR response was defined as a disappearance of HCV viral load 24 weeks after the end of the treatment.
Arm/Group | Participants With SVR | Participants Without SVR
Number analyzed (Participants) | 25 | 5
grams per liter (g/L) | -23.0 (14.768) | -32.4 (11.502)

3. Secondary Outcome: Number of Participants With Decrease in Hemoglobin
Description: The drop in hemoglobin level at Week 12 compared to level at baseline was assessed and categorized in pre-defined categories (up to 20, 20-40, greater than [>] 40 g/L) for the group of participants who achieved SVR and in the group of participants without SVR.
Time Frame: Week 12
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Participants With SVR | Participants Without SVR
Number analyzed (Participants) | 25 | 5
participants
  Up to 20 g/L | 9 | 0
  20-40 g/L | 14 | 3
  >40 g/L | 2 | 2
Statistical Analysis 1: Comparison: Participants With SVR vs Participants Without SVR; Test type: Superiority or Other; p = 0.0867, Fisher Exact

4. Secondary Outcome: Lowest Hemoglobin Level During Treatment Among Participants With or Without SVR
Description: The mean minimum hemoglobin value achieved during the treatment was assessed in the group of participants who achieved SVR and in the group of participants without SVR.
Time Frame: Week 12
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Participants With SVR | Participants Without SVR
Number analyzed (Participants) | 25 | 5
g/L | 124.24 (10.080) | 126.60 (10.383)

5. Secondary Outcome: Number of Participants With Reduction in Ribavirin Dose Due to Drop in Hemoglobin Among Participants With or Without SVR
Time Frame: Week 12
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Participants With SVR | Participants Without SVR
Number analyzed (Participants) | 25 | 5
participants | 1 | 0
Statistical Analysis 1: Comparison: Participants With SVR vs Participants Without SVR; Test type: Superiority or Other; p = 0.6492, ANCOVA

6. Secondary Outcome: Number of Participants With Neutropenia Among Participants With or Without SVR
Time Frame: Week 12
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Participants With SVR | Participants Without SVR
Number analyzed (Participants) | 25 | 5
participants | 0 | 0

7. Secondary Outcome: Number of Participants With Thrombocytopenia Among Participants With or Without SVR
Time Frame: Week 12
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Participants With SVR | Participants Without SVR
Number analyzed (Participants) | 25 | 5
participants | 1 | 0
Statistical Analysis 1: Comparison: Participants With SVR vs Participants Without SVR; Test type: Superiority or Other; p = 0.0333, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From baseline up to 24 weeks after end of treatment (up to 72 weeks)
Arm/Group | Peginterferon Alpha-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 19/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alpha-2a + Ribavirin (N=30)
Fatigue (General disorders) | 5
Influenza like illness (General disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.